CLINICAL TRIAL: NCT07335757
Title: Correlation Between C-Reactive Protein to Albumin Ratio (CAR) and Acute Kidney Injury in Patients With Acute Pancreatitis in Assiut University Hospitals.
Brief Title: C-reactive Protein & Albumin Ratio IN AKI
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Noha Fathy Radwan Abd El Zaher, dr, Assiut University
Other Study IDs: CRP and AKI
Record Dates: First submitted 2026-01-02; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Acute Kidney Injuries
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: C-reactive protein to albumin ratio — Correlation between C-Reactive Protein to Albumin Ratio (CAR) and Acute Kidney Injury in Patients with Acute Pancreatitis

SUMMARY:
Acute pancreatitis (AP), defined as acute inflammation of the pancreas, it's one of the most common diseases of the gastrointestinal tract leading to hospital admission.(1) The global incidence of AP is reported between 20 and 40 cases per 100,000 individuals, with an increasing trend over recent decades. (2) Its severity ranges from mild self-limited disease to severe acute necrotizing pancreatitis characterized by systemic complications and multi-organ failure. AKI is a frequent complication of severe acute pancreatitis, usually after the failure of other organs. (3) The aetiology of AP can be readily established in most patients. The most common causes include gallstones (40%-70%) and alcohol (25%-35%), medications as 6-mercaptopurine and azathioprine clearly can cause AP, infectious agents, and metabolic causes such as hypercalcemia and hypertriglyceridemia are rare causes (4) Acute kidney injury (AKI), affects approximately 15% of AP patients increasing to 69% in severe AP cases. AKI not only worsens the clinical status of AP patients but also significantly increases mortality risk and the likelihood of progressing to chronic kidney disease (CKD. Therefore, the challenge of early AKI identification and timely therapeutic intervention in AP patients remains critical. (2) Albumin (ALB), a negative acute-phase reactant synthesized by the liver, constitutes 40% to 60% of total plasma protein and decreases during inflammation. (5) Serum CRP refers to a positive acute phase reactant synthesized by the liver and its level in the blood elevates within hours as a response to inflammation and infection and it can be applied in follow-up owing to the short half-life, easy measurement, as well as the close association with prognosis of the disease. (6) We aimed to assess the Correlation between C-Reactive Protein to Albumin Ratio (CAR) and Acute Kidney Injury (AKI) in Patients with Acute Pancreatitis (AP) as a cost-effective, easily accessible, and reproducible prognostic biomarkers for inflammation obtained from standard blood tests.

ELIGIBILITY:
Inclusion Criteria:

* 1)patients who were diagnosed with Acute Pancreatitis by the following criteria: (i) abdominal pain mostly referred to the back, (ii) serum amylase and/or lipase greater than 3 times the upper limit of normal, and/or (iii) diagnostic findings from imaging (CT abdomen). 2)patients over 18 years old.

Exclusion Criteria:

1) Pregnant or breastfeeding women 2)Length of hospital stay ≤ 24 h 3) Patients with CKD or end-stage renal disease. 4)patients with active malignancy. 5)patients with liver cirrhosis. 6)patients with active infections or surgeries

-

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: patients with acute pancreatitis
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2029-01-30 (Estimated); Study Completion 2029-01-30 (Estimated)

PRIMARY OUTCOMES:
assessment of correlation between CRP/Alb ratio (CAR) and AKI in patients with acute pancreatitis (AP). | 10 days

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Wu W, Zhang YP, Pan YM, He ZJ, Tan YP, Wang DD, Qu XG, Zhang ZH. Predictive Value of C-Reactive Protein/Albumin Ratio for Acute Kidney Injury in Patients with Acute Pancreatitis. J Inflamm Res. 2024 Aug 16;17:5495-5507. doi: 10.2147/JIR.S473466. eCollection 2024. PMID 39165324
- [Result] Tenner S, Vege SS, Sheth SG, Sauer B, Yang A, Conwell DL, Yadlapati RH, Gardner TB. American College of Gastroenterology Guidelines: Management of Acute Pancreatitis. Am J Gastroenterol. 2024 Mar 1;119(3):419-437. doi: 10.14309/ajg.0000000000002645. Epub 2023 Nov 7. PMID 38857482